CLINICAL TRIAL: NCT00150761
Title: A Randomized, Double-blind, Double Dummy, Placebo Controlled, Cross-over Exploratory Trial in Healthy Male Adult Subjects: Comparison by Means of Infrared Thermography of the Anti-H1 Potency of Levocetirizine 5 mg and Cetirizine 10 mg Tablet Single Oral Dose After Nasal Histamine Provocation.
Brief Title: Facial Thermography Study of Levocetirizine Versus Cetirizine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: A00380
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2009-09

CONDITIONS: Anti-allergic Agents
Keywords: Nasal histamine provocation, facial thermography, levocetirizine, cetirizine,; Xyzal, Zyrtec
MeSH Terms: interventions — levocetirizine; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Levocetirizine (drug)

SUMMARY:
Phase IV, human pharmacology, exploratory, randomized, 3-way (3 treatment periods) cross-over, double blind, double dummy, placebo controlled study to compare levocetirizine and cetirizine by means of IR thermography.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Caucasian subject aged between 18 and 55 years (both inclusive).
* Subject must have a positive prick test to histamine (wheal diameter ≥ 6 mm with histamine dihydrochloride (100 mg/mL) and ≤ 3 mm with diluent control).

Exclusion Criteria:

* History of allergic disease, documented or suspected, including but not limited to: asthma, whether or not considered as allergic; nocturnal cough episode suspected to be of asthma-equivalent nature (three or more consecutive nights resulting in sleep disturbances) ; allergic rhinitis, conjunctivitis or sinusitis; nasal polyposis; dermatitis of the face or neck; drug or food allergy.
* Any clinically significant vascular disease such as hyper- or hypotension, venous disorder, vasculitis etc.
* History of hot flushes and any other vasomotor disorders.
* ENT infection or Upper Respiratory Tract Infection not completely cured at least one week before inclusion.
* Any known history of laryngeal edema.
* Nasal structural abnormalities (e.g. deviation of the nasal septum…).
* Recent immunotherapy
* Skin irritants or UV exposure 48 hours before each visit.

Ages: 18 Years to 55 Years | Sex: Male
Age Groups: Adult
Enrollment: 60
Dates: Start 2004-07; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
To compare by means of infrared (IR) thermography the anti-histaminic potency of levocetirizine 5mg (single dose) and cetirizine 5mg (single dose) using a placebo as control following 2 nasal histamine provocations (NHP) performed respectively 10 minutes

SECONDARY OUTCOMES:
To assess and compare onset of action of levocetirizine 5 mg and cetirizine 10 mg
To explore predictive value of screening thermography parameters on treatment effect
To collect additional safety information on levocetizine

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma